CLINICAL TRIAL: NCT05826925
Title: Optimizing Cardiovascular Preventive Care for Women Following Hypertensive Disorders of Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Lauren Theilen, Assistant Professor, Obstetrics & Gynecology, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00151518; K23HL159316 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-04-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hypertension, Pregnancy Induced; Hypertension Complicating Pregnancy; Preeclampsia; Cardiovascular Diseases; Patient Engagement
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Cardiovascular Diseases; Patient Participation | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid (Experimental): Participants will use the decision aid in the postpartum period
  Interventions: Other: Decision aid
- Usual care (No Intervention): Participants will receive standard postpartum care

INTERVENTIONS:
Other: Decision aid — A decision aid will be developed based on qualitative data from Aim 1 and iterative refinement with input from stakeholders from Aim 2. Anticipated content includes: 1) information about cardiovascular risk following hypertensive disorders of pregnancy; 2) goal-setting exercises for blood pressure, weight management, glucose control, physical activity, and smoking cessation; 3) self-care steps to achieve management targets; 4) values clarification exercises to identify values related to cardiovascular risk management and identify priority areas for focus and improvement; and 5) discussion of how to communicate questions and goals of treatment to their provider.
  Arms: Decision aid

SUMMARY:
Cardiovascular disease is the leading cause of death among women in the United States, and women with hypertensive disorders of pregnancy have a 2-fold higher risk for cardiovascular disease later in life compared to women with uncomplicated pregnancies. This research investigates a patient-centered intervention during the postpartum period to promote engagement in cardiovascular preventive care.

DETAILED DESCRIPTION:
Current evidence demonstrates that women with hypertensive disorders of pregnancy have 2-fold higher risk for the later development of cardiovascular disease (CVD) compared to women with healthy pregnancies. CVD prevention is a high priority for women's health, as it is the leading cause of death among women in the United States. In order to improve women's cardiovascular health, interventions for cardiovascular prevention could be initiated shortly after a pregnancy complicated by a hypertensive disorder. However, patient-centered interventions to promote preventive care engagement among postpartum women are lacking. Our objective is to address current gaps in knowledge regarding needs, values, and barriers regarding cardiovascular prevention among postpartum women with hypertensive disorders of pregnancy, and to remedy the lack of available evidence-based interventions for this at-risk population. To this end, we will conduct a pilot study to demonstrate feasibility and preliminary efficacy of a patient decision aid to improve patient knowledge and self-efficacy regarding CVD prevention during the postpartum period

ELIGIBILITY:
Inclusion Criteria:

* Delivered a pregnancy complicated by a hypertensive disorder of pregnancy at the University of Utah during the current hospital admission
* Ability to speak and read English or Spanish
* Written informed consent obtained

Exclusion Criteria:

* Cardiovascular disease diagnosis (history of peripheral artery disease, stroke, or myocardial infarction)
* Impairment of cognitive function or vision that prohibits communication and/or reading the decision aid.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | 6-8 weeks postpartum
  Measured via the validated Decisional Conflict Scale. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)

SECONDARY OUTCOMES:
Decisional conflict | One month after the initial assessment
  Measured via the validated Decisional Conflict Scale. Scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No